CLINICAL TRIAL: NCT02263495
Title: A Phase II, Multicenter, Randomized Trial of Eribulin Plus Gemcitabine (EG) vs.Paclitaxel Plus Gemcitabine (PG) in Patients With HER2-Negative Metastatic Breast Cancer as First -Line Chemotherapy
Brief Title: Eribulin Plus Gemcitabine (EG) vs Paclitaxel Plus Gemcitabine (PG) in HER2-Negative Metastatic Breast Cancer
Acronym: EG_PG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Eisai Inc. (Industry); Dong-A ST Co., Ltd. (Industry); Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Principal Investigator, Kyung Hae Jung, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0857
Record Dates: First submitted 2014-10-06; First posted 2014-10-13 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Breast Cancer
Keywords: HER2-Negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; genexol-PM; eribulin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel & Gemcitabine(PG) (Active Comparator): Paclitaxel 175mg/m2 IV , Day1,every 3weeks Gemcitabine 1250mg/m2 IV ,Day1& Day8 every 3weeks
  Interventions: Drug: Paclitaxel; Drug: Gemcitabine
- Eribulin & Gemcitabine(EG) (Experimental): Eribulin 1.0 mg/m2, 2-5min iv ,Day1& Day8 every 3weeks Gemcitabine 1,000 mg/m2 ,Day1& Day8 every 3weeks
  Interventions: Drug: Eribulin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Paclitaxel — 175mg/m2 + D5W 500mL MIV over 3hrs before gemcitabine administration
  Other Names: Genexol,
  Arms: Paclitaxel & Gemcitabine(PG)
Drug: Eribulin — 1.0 mg/m2, 2-5min iv before gemcitabine (or miv with NS 100ml in max.)
  Other Names: Halaven,
  Arms: Eribulin & Gemcitabine(EG)
Drug: Gemcitabine — PG:1250mg/m2 + NS 100ml MIV over 30mins EG:1000mg/m2 + NS 100ml MIV over 30mins
  Other Names: Gemcit

SUMMARY:
Metastatic breast cancer (MBC) is an incurable disease and is needed to improve effective chemotherapy. Paclitaxel plus Gemcitabine (PG) combination chemotherapy is one of the preferred chemotherapeutic regimens for patients with MBC, and was found to be proper as a maintenance chemotherapy regimen with survival benefit and feasible toxicity profile as shown in a large phase III KCSG (Korean Cancer Study Group) study (Park Y et al. J Clin Oncol 31(14):1732, 2013).

Eribulin mesylate is a microtubule-targeting agent that showed improved overall survival benefit as monotherapy for MBC patients as a new chemotherapeutic agent after failure of anthracycline and taxane in EMBRACE study (Cortes J et. al. Lancet 377:914-923, 2011). Eribulin was also reported its promising efficacy in another randomized phase III study that demonstrated eribulin as efficacious as capecitabine (Kaufman P et. al. Abstr# S6-6, SABCS 2012). Both study results showed potential clinical benefit in patients with triple negative MBC (TNBC). Thus, eribulin combined with gemcitabine may be a new potential regimen for early line therapy in patients with metastatic breast cancer.

Furthermore, eribulin may have rational benefit compared with paclitaxel in terms of neurotoxicity. Although there is no direct evidence that eribulin has better neurotoxicity profile than taxane, eribulin tended to show less neurotoxicity compared with ixabepilone in a phase II trial (Vahdat, L et al. 2011 SABCS). Eribulin has no worsen toxicity as compared to paclitaxel. Therefore, EG may have less neurotoxicity comparing to PG.

In phase I trial, eribulin in combination with gemcitabine was feasible in patients with advanced solid tumor treated with chemotherapy (< 3 lines) (Goel R, et al, 2009 ASCO).

Based on this rationale, the investigators are to conduct randomized phase II study comparing EG chemotherapy with PG chemotherapy for patients with HER-2 negative MBC as first-line chemotherapy.

A total of 118 patients will be recruited. Patients will be randomized to a treatment arm by permutated method. The randomization ratio is 1:1. This study is multi-center, randomized, open label study.

DETAILED DESCRIPTION:
A total of enrolled 118 patients in EG and PG groups, will be provided chemotherapy regimen:

Paclitaxel/Gemcitabine (PG) : every 3 weeks D1 Paclitaxel 175mg/m2 + D5W 500mL MIV over 3hrs before gemcitabine administration D1, D8 Gemcitabine 1,250 mg/m2 + NormalSaline 100ml MIV over 30mins

* Pre & Post medication (which can be changed according to institutions' policy) D1 Corticosteroid 100 mg i.v. 30 min. before Paclitaxel Pheniramine 1A + D5W 50mL MIV 30mins before Paclitaxel Ranitidine 50mg IV + D5W 50mL MIV 30mins before Paclitaxel HT3 antagonist 1A + D5W 50 mL MIV 30mins before Paclitaxel

Eribulin/Gemcitabine (EG): every 3weeks D1, D8 Eribulin 1.0 mg/m2, 2-5min iv before gemcitabine (or miv with NormalSaline 100ml in max.) D1, D8 Gemcitabine 1000 mg/m2 + NormalSaline100ml MIV over 30mins

<schedule of Assessment adn procedures (±3 days window period ) >

1. screening /baseline

   * obtaining Informed consent form
   * collecting information
   * demographic data
   * breast cancer treatment history/ medical history
   * general physical examination/ vital sign & Performance status
   * Test: CBC/blood chemistry/ Tumor response(CT or MRI)/
   * collecting QOL questionnaire using FACT-Taxane
2. cycle 1 ~ prior to EOT

   * general physical examination/ vital sign & Performance status
   * Test: CBC/blood chemistry/ Tumor response(CT or MRI)
   * collecting QOL questionnaire using FACT-Taxane
   * administration PG or EG
3. EOT(end of treatment)

   * general physical examination/ vital sign & Performance status
   * Test: CBC/blood chemistry/ Tumor response(CT or MRI)
   * collecting QOL questionnaire using FACT-Taxane
4. survival follow up(every 12weeks)

   * survival
   * anti neoplastic therapy after end of treatment
   * The tumor response will be performed every 12 (±2) weeks until disease progression

<WITHDRAWAL OF SUBJECTS>

Subjects may be withdrawn from the study (i.e. from any further study medication or study procedure) for the following reasons:

* At their own request
* If, in the investigator's opinion, continuation in the study would be detrimental to the subject's well-being
* In case of disease progression
* In case of unacceptable toxicity

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic, or recurrent breast cancer
2. HER2-negative breast cancer
3. age > 18 years
4. ECOG performance status 0 - 2
5. Pre- or postmenopausal breast cancer patients with measurable or non-measurable lesions, who are candidates for chemotherapy
6. Life expectancy ≥ 3 months
7. No prior history of chemotherapy for metastatic, recurrent breast cancer
8. Patients may have received prior neoadjuvant or adjuvant taxane regimen as long as it has been 12 months since completion of regimen.
9. Patients either may or may not have a prior anthracycline containing regimen.
10. Prior hormonal therapy as a treatment of metastatic disease is allowed. But antitumoral hormonal therapy must be terminated prior to enrollment(up to the date of randomization)
11. Prior radiation therapy allowed as long as < 25% of the bone marrow has been treated, and the patients must have recovered from the acute toxic effects of the treatment prior to study enrollment. Prior radiation to the whole pelvis is not allowed. Prior radiotherapy must be completed 2 weeks before study entry.
12. Bisphosphonates for the treatment of bone metastases should not be initiated following the first dose of randomized therapy. It must be initiated prior to day of treatment (cycle 1, day 1). Patients may continue on bisphosphonates who already established on bisphosphonate therapy for bone metastases
13. Adequate bone marrow function (≥ ANC 1,500/ul, ≥ platelet 100,000/ul, ≥ Hemoglobin 9.0 g/dl)
14. Adequate renal function (≤ serum creatinine 1.5 mg/dl or CCr ≥ 50 ml/min)
15. Adequate liver function (≤ serum bilirubin 1.5 mg/dl, ≤ AST & ALTX3 upper normal limit or AST and ALT ≤ 5.0XULN if judged by the investigator to be related to liver metastases)
16. Written informed consent

Exclusion Criteria:

1. Serious uncontrolled intercurrent infections
2. Serious intercurrent medical or psychiatric illness, including active cardiac disease
3. Pregnancy or breast feeding
4. Second primary malignancy(except in situ carcinoma of the cervix or adequately treated nonmelanomatous carcinoma of the skin or other malignancy treated at least 5 years previously with no evidence of recurrence)
5. Documented parenchymal or leptomeningeal brain metastasis
6. Peripheral neuropathy ≥ grade 2
7. Prior treatment with gemcitabine will not be allowed.
8. HER-2 overexpressing breast cancer and concomitant trastuzumab treatment is not allowed
9. Women of childbearing potential, unwilling to use a medically acceptable method of contraception during the trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2014-12-19 (Actual); Primary Completion 2017-05-11 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 48months
  To demonstrate that EG is not inferior to PG group in terms of PFS in patients with metastatic or recurrent breast cancer as first-line treatment.

SECONDARY OUTCOMES:
overall survival | 48months
  Survival will be measured as the time from randomization to the date of death.
neuropathic scale | expected at 9week , expected at 24week
  FACT for Taxane QOL assessment
toxicity of study drugs | from first administration until 28 days after the last dose administration
  Using CTCAE Version 4.0
duration of response | 48months
  using RECIEST version 1.1
objective response rate | 48months
  using RECIEST version 1.1
clinical benefit rate | 48months
  using RECIEST version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hae Jung, Dr, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul

REFERENCES:
- [Derived] Kim JY, Lee E, Park K, Im SA, Sohn J, Lee KS, Chae YS, Kim JH, Kim TY, Jung KH, Park YH; Breast Cancer Committee of the Korean Cancer Study Group. Exploratory biomarker analysis from a phase II clinical trial of eribulin plus gemcitabine versus paclitaxel plus gemcitabine for HER2-negative metastatic breast cancer patients (KCSG BR13-11). Breast Cancer Res Treat. 2019 Nov;178(2):367-377. doi: 10.1007/s10549-019-05400-y. Epub 2019 Aug 12. PMID 31407230
- [Derived] Park YH, Im SA, Kim SB, Sohn JH, Lee KS, Chae YS, Lee KH, Kim JH, Im YH, Kim JY, Kim TY, Lee KH, Ahn JH, Kim GM, Park IH, Lee SJ, Han HS, Kim SH, Jung KH; Korean Cancer Study Group (KCSG). Phase II, multicentre, randomised trial of eribulin plus gemcitabine versus paclitaxel plus gemcitabine as first-line chemotherapy in patients with HER2-negative metastatic breast cancer. Eur J Cancer. 2017 Nov;86:385-393. doi: 10.1016/j.ejca.2017.10.002. Epub 2017 Nov 5. PMID 29100193